CLINICAL TRIAL: NCT02475798
Title: Clinical Study to Collect Confirmatory Safety and Effectiveness of the Zenith® Branch Endovascular Graft-Iliac Bifurcation
Brief Title: PRESERVE-Zenith® Branch Endovascular Graft-Iliac Bifurcation
Status: No longer available | Type: Expanded Access
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 05-625 CA-P2
Record Dates: First submitted 2015-06-15; First posted 2015-06-19 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Aortoiliac Aneurysms; Iliac Aneurysms
Keywords: Zenith aortoiliac aneurysm; Iliac aneurysm; Branch; Connections; Endovascular graft; Graft-iliac bifurcation; Aneurysm; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Iliac Aneurysm; Aneurysm; Vascular Diseases; Cardiovascular Diseases

INTERVENTIONS:
Device: Zenith® Branch Endovascular Graft-Iliac Bifurcation, — Implantation of the following devices: Zenith® Branch Endovascular Graft-Iliac Bifurcation, the Atrium iCAST™, and the Zenith® Flex AAA Endovascular Graft.
  Other Names: Branch Graft

SUMMARY:
The purpose of this extended study is to collect confirmatory safety and effectiveness data on the Zenith® Branch Endovascular Graft-Iliac Bifurcation in combination with the commercially available Atrium iCAST™ covered stent in the treatment of aortoiliac and iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* An aortoiliac or iliac aneurysm of appropriate size
* Unsuitable distal sealing site for a traditional Zenith® iliac leg graft within the common iliac artery

Exclusion Criteria:

* Less than 18 years of age
* Inability or refusal to give informed consent
* Disease considerations that would compromise patient safety or study outcomes
* Unsuitable arterial anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: W. Anthony Lee, MD, Principal Investigator — Christine E. Lynn Heart and Vascular Institute
Locations (26):
- United States (26):
  - Mayo Foundation for Medical Education and Research, Phoenix, Arizona
  - VA Palo Alto HCS, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - Christine E. Lynn Heart and Vascular Institute, Boca Raton, Florida
  - South Florida Medical Imaging, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - St. Anthony's Medical Center, Rockford, Illinois
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Massachusetts, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital East Communities, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Aurora St. Luke's Hospital, Milwaukee, Wisconsin